CLINICAL TRIAL: NCT01251679
Title: Study to Assess Effectiveness of Nonpharmaceutical Interventions (Handwashing, Face Mask Use) to Prevent Influenza Transmission in Households
Brief Title: Household Influenza Transmission Study
Acronym: HITS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Ministry of Health, Thailand (Other Government); Armed Forces Research Institute of Medical Sciences, Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CDC-NCIRD-5288
Record Dates: First submitted 2010-12-01; First posted 2010-12-02 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Influenza
Keywords: handwashing; masks; infectious disease transmission
MeSH Terms: conditions — Influenza, Human | interventions — Hand Disinfection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (No Intervention): Control: nutrition, physical activity and smoking cessation education
- Hand washing (Experimental): Intervention 1: hand washing education and material
  Interventions: Behavioral: Hand washing
- Hand washing and surgical mask (Experimental): Intervention 2: hand washing education and material AND paper surgical face masks
  Interventions: Device: Hand washing and surgical mask

INTERVENTIONS:
Behavioral: Hand washing — hand washing education and material
  Arms: Hand washing
Device: Hand washing and surgical mask — hand washing education and material and paper surgical face masks
  Arms: Hand washing and surgical mask

SUMMARY:
The purpose of this study is to determine whether nonpharmaceutical interventions (i.e., handwashing and masks) reduce secondary transmission of influenza in households.

DETAILED DESCRIPTION:
HITS is a multi-year project that will prospectively identify laboratory-confirmed influenza infected children. Secondary influenza infection will then be examined among members of the child's household and effectiveness of non-pharmaceutical interventions to decrease secondary infection will be assessed. The pediatric influenza-infected index case will be identified by rapid influenza testing and their household will then be enrolled and randomized to one of three study arms: control, hand washing (Intervention 1), and hand washing and mask use (Intervention 2). Following enrollment, at days 0, 3 and 7, all household participants will be tested: the index case will be assessed for influenza viral shedding and household members will be assessed for secondary influenza infection. This study is being conducted at Queen Sirikit Institute for Child Health in Bangkok.

ELIGIBILITY:
Inclusion Criteria:

* Child, 1 month through 15 years of age
* Resident of Bangkok Metropolitan Area
* Outpatient of Queen Sirikit National Institute of Child Health Children's
* Hospital seen during HITS' active study period
* Positive influenza rapid test result from patient presenting with influenza-like illness
* In addition to the index case, consent must be obtained from at least 2 household members ≥1 month of age who plan to sleep inside the house for a period of at least 21 days from the time of enrollment

Exclusion Criteria:

* Illness onset 48 hours or more before presentation and influenza testing at Queen Sirikit National Institute of Child Health Children's Hospital
* Treatment with influenza antiviral medications since it may decrease secondary attack rate
* Children who are at high risk for severe influenza disease (e.g., chronic lung disease, renal disease, chemotherapy for cancer, long-term aspirin therapy)
* A history of influenza-like illness in another household member that precedes the index case by 7 days or less will lead to exclusion of the household because the source of influenza infection for secondary cases is uncertain.
* Receipt of influenza vaccine by any household member during the preceding 12 months.
* Prior participation in HITS.

Ages: 1 Month to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2920 (Actual)
Dates: Start 2008-04-09 (Actual); Primary Completion 2012-11-12 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Secondary influenza infection in household members | 21 days
  To determine the secondary attack rate (SAR) in households with a child with laboratory-confirmed influenza infection.

CONTACTS AND LOCATIONS:
Overall Officials: Sonja J Olsen, PhD, Principal Investigator — Centers for Disease Control and Prevention
Locations (1):
- Queen Sirikit National Institute of Child Health, Ratchathewi, Bangkok, Thailand

REFERENCES:
- [Result] Simmerman JM, Suntarattiwong P, Levy J, Gibbons RV, Cruz C, Shaman J, Jarman RG, Chotpitayasunondh T. Influenza virus contamination of common household surfaces during the 2009 influenza A (H1N1) pandemic in Bangkok, Thailand: implications for contact transmission. Clin Infect Dis. 2010 Nov 1;51(9):1053-61. doi: 10.1086/656581. PMID 20879867
- [Result] Suntarattiwong P, Jarman RG, Levy J, Baggett HC, Gibbons RV, Chotpitayasunondh T, Simmerman JM. Clinical performance of a rapid influenza test and comparison of nasal versus throat swabs to detect 2009 pandemic influenza A (H1N1) infection in Thai children. Pediatr Infect Dis J. 2010 Apr;29(4):366-7. doi: 10.1097/INF.0b013e3181c6f05c. PMID 19949356